CLINICAL TRIAL: NCT02581046
Title: Effect of the Timing of Lens-removal Cataract Surgery on Postoperative Complications Rate Among Patients With Bilateral Congenital Cataracts
Brief Title: Effect of the Timing of Cataract Surgery on Complications in Patients With Bilateral Congenital Cataracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Principal Investigator, Haotian Lin, Childhood Cataract Program of the Chinese Ministry of Health(CCPMOH), Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCPMOH2010-China7
Record Dates: First submitted 2015-10-16; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3 month surgical group (Experimental): Phacoemulsification pediatric cataract surgery is performed at the age of 3 month of patients without IOL implantation.
  Interventions: Procedure: Phacomulsification lens removal cataract surgery without Intraocular lens(IOL) implantation at the age of 3month of the patients; Drug: Subconjunctival dexamethasone and general anesthesia
- 6 month surgical group (Experimental): Phacoemulsification pediatric cataract surgery is performed at the age of 3 month of patients without IOL implantation..
  Interventions: Procedure: Phacomulsification lens removal cataract surgery without Intraocular lens(IOL) implantation at the age of 6 month of the patients; Drug: Subconjunctival dexamethasone and general anesthesia

INTERVENTIONS:
Procedure: Phacomulsification lens removal cataract surgery without Intraocular lens(IOL) implantation at the age of 3month of the patients — The surgical timing of phacoemulsification is perform at the age of 3 month of the patients. During Phacoemulsification, viscoelastic materials and anterior lens capsule are used to protect corneal endothelial cells.
  Arms: 3 month surgical group
Procedure: Phacomulsification lens removal cataract surgery without Intraocular lens(IOL) implantation at the age of 6 month of the patients — The surgical timing of phacoemulsification is perform at the age of 6 month of the patients. During Phacoemulsification, viscoelastic materials and anterior lens capsule are used to protect corneal endothelial cells.
  Arms: 6 month surgical group
Drug: Subconjunctival dexamethasone and general anesthesia — All patients received subconjunctival dexamethasone (2 mg) during surgery, and all surgeries were performed under general anesthesia.

SUMMARY:
Congenital cataract is an important treatable cause of visual handicap in childhood throughout the world. Successful management of childhood cataract is dependent on individualized treatment strategies and rigorous postoperative supervision for adverse complication. In this trial, we aimed to compare the difference of postoperative outcome between surgical timing at age of 3 month and 6 month. Patients enrolled into the study will be followed for two year and will have study visits at 1 day, 1 week, 1 month, 3 month, 6 month, 9 month, 12 month, 18month and 24month postoperatively.

DETAILED DESCRIPTION:
Congenital cataract is a priority of Vision 2020: the Right to Sight, the global initiative to reduce the world's burden of avoidable blindness, because it is an important treatable cause of visual handicap in childhood throughout the world. Successful management of childhood cataract is dependent on individualized treatment strategies and postoperative supervision for adverse complication is also essential. The timing of surgery of childhood cataract depends on the etiology and on the degree of visual interference. Severe bilateral cataracts with significant obstruction of the visual axis must be treated and surgery is recommended as soon as possible after discovery.

Several previous studies claimed that ideally cataracts should be removed before 3 months of age, while the result of recent researches shows that too early intervention for cataract surgery seems aggressive and would cause serious complications, which might cause poor long-term visual outcomes. Therefore, in order to control childhood blindness and severe visual impairment in China, it is of great importance to ensure that pediatric patients with cataract could have good timing of surgery, postoperative rigorous supervision, accurate optical rehabilitation and comprehensive treatment of amblyopia.

In this trial, we aimed to compare the difference of postoperative outcome between surgical timing at age of 3 month and 6 month. Patients enrolled into the study will be followed for two year and will have study visits at 1 day, 1 week, 1 month, 3 months, 6 months, 9 months, 12 months, 18months and 24months after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosis with bilateral congenital cataract for entire lens without other ocular abnormality
* No more than 3 month old
* Have signed a consent form
* Can be followed

Exclusion Criteria:

* Children not identified with congenital cataract
* Have not signed consent form
* Be not able to be followed

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the central subfield thickness (CST) measured by Optical Coherence Tomography(OCT) | during surgery,postoperation time:1day,1week,1month,3month,6month,9month,12month,18month,24month
Change from baseline in the thickness of the inner retinal layer regions measured by Optical Coherence Tomography(OCT) | during surgery,postoperation time:1day,1week,1month,3month,6month,9month,12month,18month,24month
Change from baseline in the thickness of the outer retinal layer regions measured by Optical Coherence Tomography(OCT) | during surgery,postoperation time:1day,1week,1month,3month,6month,9month,12month,18month,24month

SECONDARY OUTCOMES:
Number of participants with abnormal intraocular pressure or diagnosis with secondary glaucoma | 2 year after surgery
Number of participants undergoing Nd:YAG laser capsulotomy due to severe posterior capsular opacification（PCO） | 2 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yizhi Liu, M.D., Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University; Weirong Chen, M.D., Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zetterstrom C, Lundvall A, Kugelberg M. Cataracts in children. J Cataract Refract Surg. 2005 Apr;31(4):824-40. doi: 10.1016/j.jcrs.2005.01.012. PMID 15899463
- [Background] Whitman MC, Vanderveen DK. Complications of pediatric cataract surgery. Semin Ophthalmol. 2014 Sep-Nov;29(5-6):414-20. doi: 10.3109/08820538.2014.959192. PMID 25325868
- [Background] Mansouri B, Stacy RC, Kruger J, Cestari DM. Deprivation amblyopia and congenital hereditary cataract. Semin Ophthalmol. 2013 Sep-Nov;28(5-6):321-6. doi: 10.3109/08820538.2013.825289. PMID 24138041
- [Background] Lenhart PD, Courtright P, Wilson ME, Lewallen S, Taylor DS, Ventura MC, Bowman R, Woodward L, Ditta LC, Kruger S, Haddad D, El Shakankiri N, Rai SK, Bailey T, Lambert SR. Global challenges in the management of congenital cataract: proceedings of the 4th International Congenital Cataract Symposium held on March 7, 2014, New York, New York. J AAPOS. 2015 Apr;19(2):e1-8. doi: 10.1016/j.jaapos.2015.01.013. PMID 25892047
- [Background] Magli A, Forte R, Rombetto L. Long-term outcome of primary versus secondary intraocular lens implantation after simultaneous removal of bilateral congenital cataract. Graefes Arch Clin Exp Ophthalmol. 2013 Jan;251(1):309-14. doi: 10.1007/s00417-012-1979-7. Epub 2012 Mar 14. PMID 22411128
- [Background] Young MP, Heidary G, VanderVeen DK. Relationship between the timing of cataract surgery and development of nystagmus in patients with bilateral infantile cataracts. J AAPOS. 2012 Dec;16(6):554-7. doi: 10.1016/j.jaapos.2012.08.008. PMID 23237753
- [Background] Bayoumi NH. Surgical Management of Glaucoma After Congenital Cataract Surgery. J Pediatr Ophthalmol Strabismus. 2015 Jul-Aug;52(4):213-20. doi: 10.3928/01913913-20150414-11. Epub 2015 Apr 17. PMID 25915009
- See also: Home page of Zhongshan Ophthalmic Center — http://www.gzzoc.com/
- See also: Homepage of Childhood Cataract Program of the Chinese Ministry of Health(CCPMOH) — http://www.cnccclub.com/